CLINICAL TRIAL: NCT01996605
Title: Efficacy of Intrathecal Oxytocin in Human Volunteers
Brief Title: Efficacy of Spinal Oxytocin in Healthy Volunteers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Cessation of funding period prior to completion, due to slow recruitment during the pandemic
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00025901
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Results first posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2022-11

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Subjects are randomized into one of 3 groups to receive, in a double-blind manner, intrathecal saline or intrathecal oxytocin, 15 mcg or 150 mcg
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization is prepared by a statistician not otherwise involved in the study or data analysis and is maintained by the Wake Forest University School of Medicine research pharmacy. Study drug is dispensed by the research pharmacy labelled as "Study drug containing normal saline or oxytocin 15 mcg in normal saline or oxytocin 150 mcg in normal saline" to indicate the possible contents of the solution, thereby maintaining blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Oxytocin 15 mcg (Experimental): Oxytocin 15 mcg injected spinally
  Interventions: Drug: Oxytocin 15 mcg
- Oxytocin 150 mcg (Experimental): Oxytocin 150 mcg injected spinally
  Interventions: Drug: Oxytocin 150 mcg
- Placebo (Active Comparator): Preservative free normal saline injected spinally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin 15 mcg — Oxytocin 15 mcg will be administered spinally
  Arms: Oxytocin 15 mcg
Drug: Oxytocin 150 mcg — Oxytocin 150 mcg will be administered spinally
  Arms: Oxytocin 150 mcg
Drug: Placebo — placebo will be administered spinally
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effect of intrathecal oxytocin on areas and intensity of hyperalgesia and allodynia induced by topical capsaicin.

DETAILED DESCRIPTION:
Purpose: There is a strong experimental basis to support the study of oxytocin by the spinal route for analgesia in humans. Oxytocin containing cells in the dorsal parvocellular division of the paraventricular nucleus (PVN) project to the spinal cord (1). Noxious stimulation activates these cells via the A1 noradrenergic relay in the pons (2) and produces analgesia by spinal release of oxytocin, since intrathecal injection of an oxytocin receptor antagonist worsens pain behaviors from peripheral inflammation (3). Direct electrical stimulation of the PVN reduces dorsal horn neuronal responses to noxious stimulation, and this is blocked by administration of sequestering antibody for oxytocin (4). Similarly, direct electrical stimulation of the PVN reduces behavioral sensitivity in a model of chronic neuropathic pain, and this effect is blocked by an oxytocin receptor antagonist (5). Intrathecal injection of oxytocin in normal rats reduces dorsal horn neuronal responses to noxious stimuli (6) as well as behavioral responses to noxious thermal (3), mechanical (3), and chemical (7) stimuli. Finally, intrathecal injection of oxytocin in rat models of chronic pain also reduces dorsal horn neuronal responses to sensory stimulation (6) as well as behavioral responses to thermal (5) and mechanical (7) stimuli.

Rationale: We anticipate that oxytocin will be effective after spinal injection in humans against chemical induced hypersensitivity states.

Objectives: Determine the effect of intrathecal oxytocin on areas and intensity of hyperalgesia and allodynia induced by topical capsaicin.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* weight < 240 pounds
* American Society of Anesthesiology Category 1 or 2

Exclusion Criteria:

* allergy to oxytocin or lidocaine
* allergy to chilli peppers
* Females: active gynecological disease such as uterine fibroids or ongoing bleeding
* Pregnancy or currently breastfeeding
* Females that have delivered a baby within 2 years of study
* Taking prescription medications (exception: oral birth control medication)

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01-02; Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C Eisenach, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from Jan 2, 2014 to Oct 9, 2018 within Wake Forest University Health Sciences (WFUHS) and the community using IRB-approved advertisements. Screening for eligibility and informed consent was obtained at the Pain Mechanisms Laboratory Clinical Research Unit of WFUHS.
Period: Overall Study
Arm/Group | Oxytocin 15 mcg | Oxytocin 150 mcg | Placebo
Started | 8 | 5 | 7
Completed | 8 | 5 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin 15 mcg | Oxytocin 150 mcg | Placebo | Total
Number analyzed (Participants) | 8 | 5 | 7 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (11) | 35 (9) | 38 (10) | 36 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 4 | 10
  Male | 3 | 4 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 5 | 6 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 3
  White | 6 | 4 | 7 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 5 | 7 | 20
Area of hyperalgesia [Mean (Standard Deviation); unit: square centimeters] — Area of hyperalgesia was determined by applying a von Frey filament to the skin with normal sensation and sequentially approaching the site of capsaicin application along a radial line until the participant indicated the sensation changed from normal to a prick or pain sensation. This point was marked and the area determined.
  NOTE: At baseline prior to capsaicin application there was no hyperalgesia, so all values are 0.
  square centimeters | 0 (0) | 0 (0) | 0 (0) | 0 (0)

OUTCOME MEASURES:

1. Primary Outcome: Hyperalgesia
Description: The area of hyperalgesia after the first skin heating following topical capsaicin.
Time Frame: 105 minutes after study drug injection
Population: Area of hyperalgesia was determined as described in baseline measures 105 min after study drug injection. The sequence of events was study drug injection followed in 30 min by 5 min heating of the skin followed by capsaicin cream application for 30 min, removal of the cream followed in 30 min by 5 min heating of the skin. After this second heating the area of hyperalgesia was measured.
Measure: Mean (Standard Deviation); unit: square centimeters
Arm/Group | Oxytocin 15 mcg | Oxytocin 150 mcg | Placebo
Number analyzed (Participants) | 8 | 5 | 7
square centimeters | 103 (55) | 102 (76) | 75 (33)
Statistical Analysis 1: Comparison: Oxytocin 15 mcg vs Oxytocin 150 mcg vs Placebo; The null hypothesis was that there would be no difference in area of hyperalgesia 105 minutes after study drug injection among the three groups; Test type: Superiority; p < 0.05, ANOVA — T; A one-way ANOVA was performed on the single primary outcome datapoint comparing the three groups

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Oxytocin 15 mcg | Oxytocin 150 mcg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/5 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/5 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/5 | 0/7

LIMITATIONS AND CAVEATS:
The study was powered for a sample size of 40 and was terminated early with a sample size of 20 due to slow recruitment and cessation of financial support.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/05/NCT01996605/Prot_SAP_001.pdf
  • Informed Consent Form (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/05/NCT01996605/ICF_000.pdf